CLINICAL TRIAL: NCT04807764
Title: Priming with High-Frequency Trans-spinal Stimulation to Augment Locomotor Benefits in Spinal Cord Injury
Brief Title: Transspinal Stimulation Plus Locomotor Training for SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York (Other)
Collaborators: Bronx Veterans Medical Research Foundation, Inc (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Maria Knikou, PT, PhD, Professor/Principal Investigator, City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD100544 (NIH)
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries; Paraplegia, Spinal; Tetraplegia/Tetraparesis; Paraplegia, Spastic
Keywords: Locomotor Training; Transcutaneous Spinal Cord Stimulation; Lokomat; Peripheral Nerve Stimulation; H-Reflex; Spinal Neural Circuits; Neuroplasticity; Recovery
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia

STUDY DESIGN:
Intervention Model Description: This is a mechanistic randomized clinical trial. We will enroll 45 individuals with SCI. We will use blocked randomization into three groups with a block size of nine, with stratification according to severity of SCI (ambulatory with assistive device, or not ambulatory).1 We will check after completion of intervention by all subjects in each group whether the groups are balanced or not regarding baseline motor function and perform tests of association accordingly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Real transspinal stimulation delivered during standing followed by locomotor training (Experimental): Transspinal tonic stimulation of the thoracolumbar region will be delivered at a frequency of 30 Hz during standing with as needed body weight support (BWS) in a standing frame or in the Lokomat to ensure safety.
  Interventions: Combination Product: Standing transspinal stimulation followed by robotic gait training
- Real transspinal stimulation delivered while lying supine followed by locomotor training (Experimental): Transspinal tonic stimulation will be delivered at a frequency of 30 Hz while lying supine.
  Interventions: Combination Product: Lying transspinal stimulation followed by robotic gait training
- Sham transspinal stimulation delivered during standing followed by locomotor training (Sham Comparator): One sham group will be receiving transspinal stimulation during standing at an intensity where sensation is absent.
  Interventions: Other: Standing sham transspinal stimulation followed by robotic gait training

INTERVENTIONS:
Combination Product: Standing transspinal stimulation followed by robotic gait training — Fifteen people with spinal cord injury will receive 40 daily sessions of 30 minutes of non-invasive high frequency (e.g. 30 Hz) transcutaneous transspinal stimulation during standing followed by 30 minutes of assisted stepping robotic gait training. Before and after training standardized clinical and neurophysiological tests will be used to assess recovery of sensorimotor function.
  Other Names: Standing transspinal stimulation
  Arms: Real transspinal stimulation delivered during standing followed by locomotor training
Combination Product: Lying transspinal stimulation followed by robotic gait training — Fifteen people with spinal cord injury will receive 40 daily sessions of 30 minutes of non-invasive high frequency (e.g. 30 Hz) transcutaneous transspinal stimulation while lying supine on a therapy table followed by 30 minutes of assisted stepping robotic gait training. Before and after training standardized clinical and neurophysiological tests will be used to assess recovery of sensorimotor function.
  Other Names: Lying transspinal stimulation
  Arms: Real transspinal stimulation delivered while lying supine followed by locomotor training
Other: Standing sham transspinal stimulation followed by robotic gait training — Fifteen people with spinal cord injury will receive 40 daily sessions of 30 minutes of sham transspinal stimulation during standing at an intensity where sensation is absent followed by 30 minutes of robotic gait training. Before and after training standardized clinical and neurophysiological tests will be used to assess recovery of sensorimotor function.
  Other Names: Robotic gait training
  Arms: Sham transspinal stimulation delivered during standing followed by locomotor training

SUMMARY:
Locomotor training is often used with the aim to improve corticospinal function and walking ability in individuals with Spinal Cord Injury. Excitingly, the benefits of locomotor training may be augmented by noninvasive electrical stimulation of the spinal cord and enhance motor recovery at SCI. This study will compare the effects of priming locomotor training with high-frequency noninvasive thoracolumbar spinal stimulation. In people with motor-incomplete SCI, a series of clinical and electrical tests of brain and spinal cord function will be performed before and after 40 sessions of locomotor training where spinal stimulation is delivered immediately before either lying down or during standing.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) greatly impairs standing and walking ability, which severely compromises daily living activities. While these deficits are partially improved by locomotor training, even after multiple training sessions, abnormal muscle activity and coordination still persist. Thus, locomotor training alone cannot fully optimize the neuronal plasticity required to strengthen the synapses connecting the brain, spinal cord, and local circuits. As such, treatment interventions that effectively promote neuromodulation of spinal locomotor networks and strengthen neural connectivity of the injured human spinal cord in combination with physical rehabilitation are greatly needed. It is proposed that transcutaneous spinal cord (transspinal) stimulation as a method to synergistically 'prime' the nervous system to better respond to locomotor training. Transspinal stimulation alters motoneuron excitability over multiple spinal segments, a pre-requisite for functioning descending and local inputs. Importantly, whether concurrent treatment with transspinal stimulation and locomotor training maximizes motor recovery after SCI is unknown. The goal of this clinical trial is to use high frequency (30 Hz) transspinal stimulation to prime locomotor training and ultimately improve standing, walking, and overall function in individuals with chronic incomplete SCI (iSCI). Forty-five individuals with iSCI will undergo 40 sessions of body weight-supported step training primed with high-frequency transspinal stimulation. Participants will be randomized to receive transspinal stimulation during standing (real or sham) or while supine (real). Aim 1 evaluates how priming locomotor training with high-frequency transspinal stimulation in SCI alters corticomotoneuronal connectivity strength, as indicated by motor evoked potentials recorded from the legs.

Aim 2 evaluates how priming locomotor training with high-frequency transspinal stimulation in iSCI affects reorganization and appropriate engagement of spinal neuronal circuits. Finally, Aim 3 evaluates activity-based motor function, ability to stand and walk, and quality of life. These results will support the notion that tonic high-frequency transspinal stimulation strengthens corticomotoneuronal connectivity and improves spinal circuit organization through posture-dependent corticospinal neuroplasticity. It is anticipated that the information gained from this mechanistic clinical trial will greatly impact clinical practice. This is because in real-world clinical settings, noninvasive transspinal stimulation can be more easily and widely implemented than invasive epidural stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with all study procedures and availability for the duration of the study.
* Ability to understand the consent form, and sign the consent form.
* Male or female, age 18-70 years old.
* In good general health as evidenced by medical history.
* Diagnosed with motor incomplete SCI (AIS C-D).
* Bone mineral density of the hip (proximal femur) T-score <3.5 SD from age- and gender-matched normative data.
* Lesion above thoracic (T) 10 to ensure absent lower motoneuron lesion.
* Presence of tendon reflexes to be able to elicit the soleus H-reflex.
* Absent permanent ankle joint contractures that prevent passive or active ankle movement because corticospinal and spinal excitability is based on the ankle angle. The ankle straps of the Lokomat require also flexible ankle joints.
* A diagnosis of first time SCI due to trauma, vascular, or orthopedic pathology.
* Time after SCI of more than 6 months.
* Stable medical condition without cardiopulmonary disease or cognitive impairment.

Exclusion Criteria:

* Supraspinal lesions.
* Significant neuropathies of the peripheral nervous system.
* Significant degenerative neurological disorders of the spine or spinal cord.
* AIS A or B.
* Presence of pressure sores.
* Advanced urinary tract infection.
* Neoplastic or vascular disorders of the spine or spinal cord.
* Participation in an ongoing research study or new rehabilitation program.
* Pregnant women or women who suspect they may be, or may become pregnant will be excluded from participation because the risks of thoracolumbar stimulation to the fetus are unknown.
* People with cochlear implants, pacemaker, implanted infusion device, and/or implanted stimulators of any type and purpose will be excluded to avoid their malfunction due to stimulation.
* People with history of seizures.
* Medical conditions that increase the possibility of seizures.
* Medications that may change the seizure threshold.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Plasticity of spinal neuronal networks | 4 years
  Neurophysiological assessments probing changes in excitatory and inhibitory spinal reflex excitability from interventions by recording amplitude modulation of the soleus H-reflex following posterior tibial and common peroneal nerves stimulation both at rest and during robotic-assisted stepping.
Plasticity of corticospinal networks | 4 years
  Neurophysiological measurements assessing changes in corticospinal excitability from the interventions by recording responses to single-pulse transcranial magnetic stimulation (TMS) at rest and during robotic-assisted stepping.

SECONDARY OUTCOMES:
Ambulatory function | 4 years
  Change in two-minute walk and 10-meter timed test.
Balance | 4 years
  Changes in BESTtest clinical assessments.
Autonomic function | 4 years
  Questionnaire assessing participants perceived changes in bowel, bladder, and sexual function

CONTACTS AND LOCATIONS:
Overall Officials: Maria Knikou, PT, PhD, Principal Investigator — Research Foundation of the City University of New York; Noam Y. Harel, MD, PhD, Principal Investigator — Bronx Veterans Medical Research Foundation
Locations (2):
- United States (2):
  - Department of Physical Therapy, Motor Control and NeuroRecovery Laboratory, Staten Island, New York
  - Veterans Affairs Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cote MP, Murray LM, Knikou M. Spinal Control of Locomotion: Individual Neurons, Their Circuits and Functions. Front Physiol. 2018 Jun 25;9:784. doi: 10.3389/fphys.2018.00784. eCollection 2018. PMID 29988534
- [Background] Ellaway PH, Catley M, Davey NJ, Kuppuswamy A, Strutton P, Frankel HL, Jamous A, Savic G. Review of physiological motor outcome measures in spinal cord injury using transcranial magnetic stimulation and spinal reflexes. J Rehabil Res Dev. 2007;44(1):69-76. doi: 10.1682/jrrd.2005.08.0140. PMID 17551860
- [Background] Wirth B, van Hedel HJ, Curt A. Ankle paresis in incomplete spinal cord injury: relation to corticospinal conductivity and ambulatory capacity. J Clin Neurophysiol. 2008 Aug;25(4):210-7. doi: 10.1097/WNP.0b013e318183f4e3. PMID 18677185
- [Background] Cirillo J, Calabro FJ, Perez MA. Impaired Organization of Paired-Pulse TMS-Induced I-Waves After Human Spinal Cord Injury. Cereb Cortex. 2016 May;26(5):2167-77. doi: 10.1093/cercor/bhv048. Epub 2015 Mar 25. PMID 25814508
- [Background] Arvanian VL, Schnell L, Lou L, Golshani R, Hunanyan A, Ghosh A, Pearse DD, Robinson JK, Schwab ME, Fawcett JW, Mendell LM. Chronic spinal hemisection in rats induces a progressive decline in transmission in uninjured fibers to motoneurons. Exp Neurol. 2009 Apr;216(2):471-80. doi: 10.1016/j.expneurol.2009.01.004. PMID 19320005
- [Background] Nielsen JB, Crone C, Hultborn H. The spinal pathophysiology of spasticity--from a basic science point of view. Acta Physiol (Oxf). 2007 Feb;189(2):171-80. doi: 10.1111/j.1748-1716.2006.01652.x. PMID 17250567
- [Background] Knikou M. Plantar cutaneous input modulates differently spinal reflexes in subjects with intact and injured spinal cord. Spinal Cord. 2007 Jan;45(1):69-77. doi: 10.1038/sj.sc.3101917. Epub 2006 Mar 14. PMID 16534501
- [Background] Knikou M, Angeli CA, Ferreira CK, Harkema SJ. Soleus H-reflex gain, threshold, and amplitude as function of body posture and load in spinal cord intact and injured subjects. Int J Neurosci. 2009;119(11):2056-73. doi: 10.1080/00207450903139747. PMID 19863261
- [Background] Knikou M, Angeli CA, Ferreira CK, Harkema SJ. Soleus H-reflex modulation during body weight support treadmill walking in spinal cord intact and injured subjects. Exp Brain Res. 2009 Mar;193(3):397-407. doi: 10.1007/s00221-008-1636-x. Epub 2008 Nov 15. PMID 19011843
- [Background] Barthelemy D, Willerslev-Olsen M, Lundell H, Biering-Sorensen F, Nielsen JB. Assessment of transmission in specific descending pathways in relation to gait and balance following spinal cord injury. Prog Brain Res. 2015;218:79-101. doi: 10.1016/bs.pbr.2014.12.012. Epub 2015 Mar 29. PMID 25890133
- [Background] Barthelemy D, Willerslev-Olsen M, Lundell H, Conway BA, Knudsen H, Biering-Sorensen F, Nielsen JB. Impaired transmission in the corticospinal tract and gait disability in spinal cord injured persons. J Neurophysiol. 2010 Aug;104(2):1167-76. doi: 10.1152/jn.00382.2010. Epub 2010 Jun 16. PMID 20554839
- [Background] James ND, McMahon SB, Field-Fote EC, Bradbury EJ. Neuromodulation in the restoration of function after spinal cord injury. Lancet Neurol. 2018 Oct;17(10):905-917. doi: 10.1016/S1474-4422(18)30287-4. Epub 2018 Sep 18. PMID 30264729
- [Background] Tansey KE, McKay WB, Kakulas BA. Restorative neurology: consideration of the new anatomy and physiology of the injured nervous system. Clin Neurol Neurosurg. 2012 Jun;114(5):436-40. doi: 10.1016/j.clineuro.2012.01.010. Epub 2012 Feb 1. PMID 22300890
- [Background] Smith AC, Mummidisetty CK, Rymer WZ, Knikou M. Locomotor training alters the behavior of flexor reflexes during walking in human spinal cord injury. J Neurophysiol. 2014 Nov 1;112(9):2164-75. doi: 10.1152/jn.00308.2014. Epub 2014 Aug 13. PMID 25122715
- [Background] Smith AC, Rymer WZ, Knikou M. Locomotor training modifies soleus monosynaptic motoneuron responses in human spinal cord injury. Exp Brain Res. 2015 Jan;233(1):89-103. doi: 10.1007/s00221-014-4094-7. Epub 2014 Sep 10. PMID 25205562
- [Background] Martinez SA, Nguyen ND, Bailey E, Doyle-Green D, Hauser HA, Handrakis JP, Knezevic S, Marett C, Weinman J, Romero AF, Santiago TM, Yang AH, Yung L, Asselin PK, Weir JP, Kornfeld SD, Bauman WA, Spungen AM, Harel NY. Multimodal cortical and subcortical exercise compared with treadmill training for spinal cord injury. PLoS One. 2018 Aug 9;13(8):e0202130. doi: 10.1371/journal.pone.0202130. eCollection 2018. PMID 30092092
- [Background] Knikou M. Functional reorganization of soleus H-reflex modulation during stepping after robotic-assisted step training in people with complete and incomplete spinal cord injury. Exp Brain Res. 2013 Jul;228(3):279-96. doi: 10.1007/s00221-013-3560-y. Epub 2013 May 25. PMID 23708757
- [Background] Dobkin BH. Spinal and supraspinal plasticity after incomplete spinal cord injury: correlations between functional magnetic resonance imaging and engaged locomotor networks. Prog Brain Res. 2000;128:99-111. doi: 10.1016/S0079-6123(00)28010-2. No abstract available. PMID 11105672
- [Background] Thomas SL, Gorassini MA. Increases in corticospinal tract function by treadmill training after incomplete spinal cord injury. J Neurophysiol. 2005 Oct;94(4):2844-55. doi: 10.1152/jn.00532.2005. Epub 2005 Jul 6. PMID 16000519
- [Background] Wernig A, Muller S, Nanassy A, Cagol E. Laufband therapy based on 'rules of spinal locomotion' is effective in spinal cord injured persons. Eur J Neurosci. 1995 Apr 1;7(4):823-9. doi: 10.1111/j.1460-9568.1995.tb00686.x. PMID 7620630
- [Background] Knikou M, Mummidisetty CK. Locomotor training improves premotoneuronal control after chronic spinal cord injury. J Neurophysiol. 2014 Jun 1;111(11):2264-75. doi: 10.1152/jn.00871.2013. Epub 2014 Mar 5. PMID 24598526
- [Background] Knikou M, Smith AC, Mummidisetty CK. Locomotor training improves reciprocal and nonreciprocal inhibitory control of soleus motoneurons in human spinal cord injury. J Neurophysiol. 2015 Apr 1;113(7):2447-60. doi: 10.1152/jn.00872.2014. Epub 2015 Jan 21. PMID 25609110
- [Background] Ramer LM, Ramer MS, Bradbury EJ. Restoring function after spinal cord injury: towards clinical translation of experimental strategies. Lancet Neurol. 2014 Dec;13(12):1241-56. doi: 10.1016/S1474-4422(14)70144-9. Epub 2014 Nov 10. PMID 25453463
- [Background] Courtine G, Gerasimenko Y, van den Brand R, Yew A, Musienko P, Zhong H, Song B, Ao Y, Ichiyama RM, Lavrov I, Roy RR, Sofroniew MV, Edgerton VR. Transformation of nonfunctional spinal circuits into functional states after the loss of brain input. Nat Neurosci. 2009 Oct;12(10):1333-42. doi: 10.1038/nn.2401. Epub 2009 Sep 20. PMID 19767747
- [Background] Angeli CA, Boakye M, Morton RA, Vogt J, Benton K, Chen Y, Ferreira CK, Harkema SJ. Recovery of Over-Ground Walking after Chronic Motor Complete Spinal Cord Injury. N Engl J Med. 2018 Sep 27;379(13):1244-1250. doi: 10.1056/NEJMoa1803588. Epub 2018 Sep 24. PMID 30247091
- [Background] Angeli CA, Edgerton VR, Gerasimenko YP, Harkema SJ. Altering spinal cord excitability enables voluntary movements after chronic complete paralysis in humans. Brain. 2014 May;137(Pt 5):1394-409. doi: 10.1093/brain/awu038. Epub 2014 Apr 8. PMID 24713270
- [Background] Gill ML, Grahn PJ, Calvert JS, Linde MB, Lavrov IA, Strommen JA, Beck LA, Sayenko DG, Van Straaten MG, Drubach DI, Veith DD, Thoreson AR, Lopez C, Gerasimenko YP, Edgerton VR, Lee KH, Zhao KD. Publisher Correction: Neuromodulation of lumbosacral spinal networks enables independent stepping after complete paraplegia. Nat Med. 2018 Dec;24(12):1942. doi: 10.1038/s41591-018-0248-7. PMID 30353100
- [Background] Harkema S, Gerasimenko Y, Hodes J, Burdick J, Angeli C, Chen Y, Ferreira C, Willhite A, Rejc E, Grossman RG, Edgerton VR. Effect of epidural stimulation of the lumbosacral spinal cord on voluntary movement, standing, and assisted stepping after motor complete paraplegia: a case study. Lancet. 2011 Jun 4;377(9781):1938-47. doi: 10.1016/S0140-6736(11)60547-3. Epub 2011 May 19. PMID 21601270
- [Background] Rejc E, Angeli C, Harkema S. Effects of Lumbosacral Spinal Cord Epidural Stimulation for Standing after Chronic Complete Paralysis in Humans. PLoS One. 2015 Jul 24;10(7):e0133998. doi: 10.1371/journal.pone.0133998. eCollection 2015. PMID 26207623
- [Background] Rejc E, Angeli CA, Bryant N, Harkema SJ. Effects of Stand and Step Training with Epidural Stimulation on Motor Function for Standing in Chronic Complete Paraplegics. J Neurotrauma. 2017 May 1;34(9):1787-1802. doi: 10.1089/neu.2016.4516. Epub 2016 Oct 5. PMID 27566051
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Hofstoetter US, Knikou M, Guertin PA, Minassian K. Probing the Human Spinal Locomotor Circuits by Phasic Step-Induced Feedback and by Tonic Electrical and Pharmacological Neuromodulation. Curr Pharm Des. 2017;23(12):1805-1820. doi: 10.2174/1381612822666161214144655. PMID 27981912
- [Background] Pulverenti TS, Islam MA, Alsalman O, Murray LM, Harel NY, Knikou M. Transspinal stimulation decreases corticospinal excitability and alters the function of spinal locomotor networks. J Neurophysiol. 2019 Dec 1;122(6):2331-2343. doi: 10.1152/jn.00554.2019. Epub 2019 Oct 2. PMID 31577515
- [Background] Donovan J, Kirshblum S. Clinical Trials in Traumatic Spinal Cord Injury. Neurotherapeutics. 2018 Jul;15(3):654-668. doi: 10.1007/s13311-018-0632-5. PMID 29736858
- [Background] James ND, Bartus K, Grist J, Bennett DL, McMahon SB, Bradbury EJ. Conduction failure following spinal cord injury: functional and anatomical changes from acute to chronic stages. J Neurosci. 2011 Dec 14;31(50):18543-55. doi: 10.1523/JNEUROSCI.4306-11.2011. PMID 22171053
- [Background] Murray LM, Knikou M. Repeated cathodal transspinal pulse and direct current stimulation modulate cortical and corticospinal excitability differently in healthy humans. Exp Brain Res. 2019 Jul;237(7):1841-1852. doi: 10.1007/s00221-019-05559-2. Epub 2019 May 11. PMID 31079235
- [Background] Knikou M. Transpinal and transcortical stimulation alter corticospinal excitability and increase spinal output. PLoS One. 2014 Jul 9;9(7):e102313. doi: 10.1371/journal.pone.0102313. eCollection 2014. PMID 25007330
- [Background] Knikou M, Murray LM. Neural interactions between transspinal evoked potentials and muscle spindle afferents in humans. J Electromyogr Kinesiol. 2018 Dec;43:174-183. doi: 10.1016/j.jelekin.2018.10.005. Epub 2018 Oct 9. PMID 30352388
- [Background] Gerasimenko Y, Gorodnichev R, Moshonkina T, Sayenko D, Gad P, Reggie Edgerton V. Transcutaneous electrical spinal-cord stimulation in humans. Ann Phys Rehabil Med. 2015 Sep;58(4):225-231. doi: 10.1016/j.rehab.2015.05.003. Epub 2015 Jul 20. PMID 26205686
- [Background] Gerasimenko YP, Lu DC, Modaber M, Zdunowski S, Gad P, Sayenko DG, Morikawa E, Haakana P, Ferguson AR, Roy RR, Edgerton VR. Noninvasive Reactivation of Motor Descending Control after Paralysis. J Neurotrauma. 2015 Dec 15;32(24):1968-80. doi: 10.1089/neu.2015.4008. Epub 2015 Aug 20. PMID 26077679
- [Background] Gorodnichev RM, Pivovarova EA, Pukhov A, Moiseev SA, Savokhin AA, Moshonkina TR, Shcherbakova NA, Kilimnik VA, Selionov VA, Kozlovskaia IB, Edgerton VR, Gerasimenko IuP. [Transcutaneous electrical stimulation of the spinal cord: non-invasive tool for activation of locomotor circuitry in human]. Fiziol Cheloveka. 2012 Mar-Apr;38(2):46-56. Russian. PMID 22679796
- [Background] Shapkova EY, Schomburg ED. Two types of motor modulation underlying human stepping evoked by spinal cord electrical stimulation (SCES). Acta Physiol Pharmacol Bulg. 2001;26(3):155-7. PMID 11695529
- [Background] Hofstoetter US, Krenn M, Danner SM, Hofer C, Kern H, McKay WB, Mayr W, Minassian K. Augmentation of Voluntary Locomotor Activity by Transcutaneous Spinal Cord Stimulation in Motor-Incomplete Spinal Cord-Injured Individuals. Artif Organs. 2015 Oct;39(10):E176-86. doi: 10.1111/aor.12615. Epub 2015 Oct 6. PMID 26450344
- [Background] Hofstoetter US, McKay WB, Tansey KE, Mayr W, Kern H, Minassian K. Modification of spasticity by transcutaneous spinal cord stimulation in individuals with incomplete spinal cord injury. J Spinal Cord Med. 2014 Mar;37(2):202-11. doi: 10.1179/2045772313Y.0000000149. Epub 2013 Nov 26. PMID 24090290
- [Background] Minassian K, Hofstoetter US. Spinal Cord Stimulation and Augmentative Control Strategies for Leg Movement after Spinal Paralysis in Humans. CNS Neurosci Ther. 2016 Apr;22(4):262-70. doi: 10.1111/cns.12530. Epub 2016 Feb 18. PMID 26890324
- [Background] Knikou M, Hajela N, Mummidisetty CK, Xiao M, Smith AC. Soleus H-reflex phase-dependent modulation is preserved during stepping within a robotic exoskeleton. Clin Neurophysiol. 2011 Jul;122(7):1396-404. doi: 10.1016/j.clinph.2010.12.044. Epub 2011 Jan 14. PMID 21237704
- [Background] Knikou M, Hajela N, Mummidisetty CK. Corticospinal excitability during walking in humans with absent and partial body weight support. Clin Neurophysiol. 2013 Dec;124(12):2431-8. doi: 10.1016/j.clinph.2013.06.004. Epub 2013 Jun 28. PMID 23810634
- [Background] Schubert M, Curt A, Jensen L, Dietz V. Corticospinal input in human gait: modulation of magnetically evoked motor responses. Exp Brain Res. 1997 Jun;115(2):234-46. doi: 10.1007/pl00005693. PMID 9224852
- [Background] Nielsen JB. Human Spinal Motor Control. Annu Rev Neurosci. 2016 Jul 8;39:81-101. doi: 10.1146/annurev-neuro-070815-013913. Epub 2016 Mar 25. PMID 27023730
- [Background] Barthelemy D, Knudsen H, Willerslev-Olsen M, Lundell H, Nielsen JB, Biering-Sorensen F. Functional implications of corticospinal tract impairment on gait after spinal cord injury. Spinal Cord. 2013 Nov;51(11):852-6. doi: 10.1038/sc.2013.84. Epub 2013 Aug 13. PMID 23939192
- [Background] Field-Fote EC, Yang JF, Basso DM, Gorassini MA. Supraspinal Control Predicts Locomotor Function and Forecasts Responsiveness to Training after Spinal Cord Injury. J Neurotrauma. 2017 May 1;34(9):1813-1825. doi: 10.1089/neu.2016.4565. Epub 2016 Dec 20. PMID 27673569
- [Background] Zewdie ET, Roy FD, Yang JF, Gorassini MA. Facilitation of descending excitatory and spinal inhibitory networks from training of endurance and precision walking in participants with incomplete spinal cord injury. Prog Brain Res. 2015;218:127-55. doi: 10.1016/bs.pbr.2014.12.005. Epub 2015 Mar 29. PMID 25890135
- [Background] Petersen JA, Spiess M, Curt A, Dietz V, Schubert M; EM-SCI Study Group. Spinal cord injury: one-year evolution of motor-evoked potentials and recovery of leg motor function in 255 patients. Neurorehabil Neural Repair. 2012 Oct;26(8):939-48. doi: 10.1177/1545968312438437. Epub 2012 Mar 28. PMID 22460611
- [Background] Harkema SJ, Hurley SL, Patel UK, Requejo PS, Dobkin BH, Edgerton VR. Human lumbosacral spinal cord interprets loading during stepping. J Neurophysiol. 1997 Feb;77(2):797-811. doi: 10.1152/jn.1997.77.2.797. PMID 9065851
- [Background] Knikou M, Conway BA. Modulation of soleus H-reflex following ipsilateral mechanical loading of the sole of the foot in normal and complete spinal cord injured humans. Neurosci Lett. 2001 May 4;303(2):107-10. doi: 10.1016/s0304-3940(01)01718-9. PMID 11311504
- [Background] Slawinska U, Majczynski H, Dai Y, Jordan LM. The upright posture improves plantar stepping and alters responses to serotonergic drugs in spinal rats. J Physiol. 2012 Apr 1;590(7):1721-36. doi: 10.1113/jphysiol.2011.224931. Epub 2012 Feb 20. PMID 22351637
- [Background] Knikou M. Neural control of locomotion and training-induced plasticity after spinal and cerebral lesions. Clin Neurophysiol. 2010 Oct;121(10):1655-68. doi: 10.1016/j.clinph.2010.01.039. Epub 2010 Apr 27. PMID 20427232
- [Background] Rossignol S, Dubuc R, Gossard JP. Dynamic sensorimotor interactions in locomotion. Physiol Rev. 2006 Jan;86(1):89-154. doi: 10.1152/physrev.00028.2005. PMID 16371596
- [Background] Cote MP, Murray M, Lemay MA. Rehabilitation Strategies after Spinal Cord Injury: Inquiry into the Mechanisms of Success and Failure. J Neurotrauma. 2017 May 15;34(10):1841-1857. doi: 10.1089/neu.2016.4577. Epub 2016 Nov 21. PMID 27762657
- [Background] Calancie B, Broton JG, Klose KJ, Traad M, Difini J, Ayyar DR. Evidence that alterations in presynaptic inhibition contribute to segmental hypo- and hyperexcitability after spinal cord injury in man. Electroencephalogr Clin Neurophysiol. 1993 Jun;89(3):177-86. doi: 10.1016/0168-5597(93)90131-8. PMID 7686850
- [Background] Lee JK, Emch GS, Johnson CS, Wrathall JR. Effect of spinal cord injury severity on alterations of the H-reflex. Exp Neurol. 2005 Dec;196(2):430-40. doi: 10.1016/j.expneurol.2005.08.018. Epub 2005 Sep 26. PMID 16185689
- [Background] Crone C, Johnsen LL, Biering-Sorensen F, Nielsen JB. Appearance of reciprocal facilitation of ankle extensors from ankle flexors in patients with stroke or spinal cord injury. Brain. 2003 Feb;126(Pt 2):495-507. doi: 10.1093/brain/awg036. PMID 12538415
- [Background] Norton JA, Gorassini MA. Changes in cortically related intermuscular coherence accompanying improvements in locomotor skills in incomplete spinal cord injury. J Neurophysiol. 2006 Apr;95(4):2580-9. doi: 10.1152/jn.01289.2005. Epub 2006 Jan 11. PMID 16407422
- [Background] Minassian K, Hofstoetter US, Dzeladini F, Guertin PA, Ijspeert A. The Human Central Pattern Generator for Locomotion: Does It Exist and Contribute to Walking? Neuroscientist. 2017 Dec;23(6):649-663. doi: 10.1177/1073858417699790. Epub 2017 Mar 28. PMID 28351197
- [Background] Deliagina TG, Zelenin PV, Orlovsky GN. Physiological and circuit mechanisms of postural control. Curr Opin Neurobiol. 2012 Aug;22(4):646-52. doi: 10.1016/j.conb.2012.03.002. Epub 2012 Mar 23. PMID 22446009
- [Background] Horak FB, Nashner LM. Central programming of postural movements: adaptation to altered support-surface configurations. J Neurophysiol. 1986 Jun;55(6):1369-81. doi: 10.1152/jn.1986.55.6.1369. PMID 3734861
- [Background] Milosevic M, Gagnon DH, Gourdou P, Nakazawa K. Postural regulatory strategies during quiet sitting are affected in individuals with thoracic spinal cord injury. Gait Posture. 2017 Oct;58:446-452. doi: 10.1016/j.gaitpost.2017.08.032. Epub 2017 Aug 31. PMID 28910658
- [Background] Milosevic M, Yokoyama H, Grangeon M, Masani K, Popovic MR, Nakazawa K, Gagnon DH. Muscle synergies reveal impaired trunk muscle coordination strategies in individuals with thoracic spinal cord injury. J Electromyogr Kinesiol. 2017 Oct;36:40-48. doi: 10.1016/j.jelekin.2017.06.007. Epub 2017 Jul 1. PMID 28734171
- [Background] Milosevic M, Masani K, Kuipers MJ, Rahouni H, Verrier MC, McConville KM, Popovic MR. Trunk control impairment is responsible for postural instability during quiet sitting in individuals with cervical spinal cord injury. Clin Biomech (Bristol). 2015 Jun;30(5):507-12. doi: 10.1016/j.clinbiomech.2015.03.002. Epub 2015 Mar 14. PMID 25812727
- [Background] Lemay JF, Duclos C, Nadeau S, Gagnon DH. Postural control during gait initiation and termination of adults with incomplete spinal cord injury. Hum Mov Sci. 2015 Jun;41:20-31. doi: 10.1016/j.humov.2015.02.003. Epub 2015 Feb 26. PMID 25725378
- [Background] Chen YS, Zhou S. Soleus H-reflex and its relation to static postural control. Gait Posture. 2011 Feb;33(2):169-78. doi: 10.1016/j.gaitpost.2010.12.008. Epub 2011 Jan 5. PMID 21211976
- [Background] Kawaishi Y, Domen K. The relationship between dynamic balancing ability and posture-related modulation of the soleus H-reflex. J Electromyogr Kinesiol. 2016 Feb;26:120-4. doi: 10.1016/j.jelekin.2015.11.010. Epub 2015 Dec 12. PMID 26724819
- [Background] Papegaaij S, Baudry S, Negyesi J, Taube W, Hortobagyi T. Intracortical inhibition in the soleus muscle is reduced during the control of upright standing in both young and old adults. Eur J Appl Physiol. 2016 May;116(5):959-67. doi: 10.1007/s00421-016-3354-6. Epub 2016 Mar 22. PMID 27002819
- [Background] Soto O, Valls-Sole J, Shanahan P, Rothwell J. Reduction of intracortical inhibition in soleus muscle during postural activity. J Neurophysiol. 2006 Oct;96(4):1711-7. doi: 10.1152/jn.00133.2006. Epub 2006 Jun 21. PMID 16790603
- [Background] Baudry S, Penzer F, Duchateau J. Input-output characteristics of soleus homonymous Ia afferents and corticospinal pathways during upright standing differ between young and elderly adults. Acta Physiol (Oxf). 2014 Mar;210(3):667-77. doi: 10.1111/apha.12233. PMID 24433254
- [Background] Tokuno CD, Taube W, Cresswell AG. An enhanced level of motor cortical excitability during the control of human standing. Acta Physiol (Oxf). 2009 Mar;195(3):385-95. doi: 10.1111/j.1748-1716.2008.01898.x. Epub 2008 Sep 4. PMID 18774948
- [Background] Rath M, Vette AH, Ramasubramaniam S, Li K, Burdick J, Edgerton VR, Gerasimenko YP, Sayenko DG. Trunk Stability Enabled by Noninvasive Spinal Electrical Stimulation after Spinal Cord Injury. J Neurotrauma. 2018 Nov 1;35(21):2540-2553. doi: 10.1089/neu.2017.5584. Epub 2018 Jul 5. PMID 29786465
- [Background] Sayenko DG, Rath M, Ferguson AR, Burdick JW, Havton LA, Edgerton VR, Gerasimenko YP. Self-Assisted Standing Enabled by Non-Invasive Spinal Stimulation after Spinal Cord Injury. J Neurotrauma. 2019 May 1;36(9):1435-1450. doi: 10.1089/neu.2018.5956. Epub 2018 Dec 15. PMID 30362876
- [Background] Gerasimenko Y, Sayenko D, Gad P, Kozesnik J, Moshonkina T, Grishin A, Pukhov A, Moiseev S, Gorodnichev R, Selionov V, Kozlovskaya I, Edgerton VR. Electrical Spinal Stimulation, and Imagining of Lower Limb Movements to Modulate Brain-Spinal Connectomes That Control Locomotor-Like Behavior. Front Physiol. 2018 Sep 19;9:1196. doi: 10.3389/fphys.2018.01196. eCollection 2018. PMID 30283341
- [Background] Kumru H, Benito-Penalva J, Valls-Sole J, Murillo N, Tormos JM, Flores C, Vidal J. Placebo-controlled study of rTMS combined with Lokomat(R) gait training for treatment in subjects with motor incomplete spinal cord injury. Exp Brain Res. 2016 Dec;234(12):3447-3455. doi: 10.1007/s00221-016-4739-9. Epub 2016 Jul 28. PMID 27469242
- [Background] Raithatha R, Carrico C, Powell ES, Westgate PM, Chelette Ii KC, Lee K, Dunsmore L, Salles S, Sawaki L. Non-invasive brain stimulation and robot-assisted gait training after incomplete spinal cord injury: A randomized pilot study. NeuroRehabilitation. 2016;38(1):15-25. doi: 10.3233/NRE-151291. PMID 26889794
- [Background] Estes SP, Iddings JA, Field-Fote EC. Priming Neural Circuits to Modulate Spinal Reflex Excitability. Front Neurol. 2017 Feb 3;8:17. doi: 10.3389/fneur.2017.00017. eCollection 2017. PMID 28217104
- [Background] Murray LM, Knikou M. Remodeling Brain Activity by Repetitive Cervicothoracic Transspinal Stimulation after Human Spinal Cord Injury. Front Neurol. 2017 Feb 20;8:50. doi: 10.3389/fneur.2017.00050. eCollection 2017. PMID 28265259
- [Background] Knikou M, Murray LM. Repeated transspinal stimulation decreases soleus H-reflex excitability and restores spinal inhibition in human spinal cord injury. PLoS One. 2019 Sep 26;14(9):e0223135. doi: 10.1371/journal.pone.0223135. eCollection 2019. PMID 31557238
- [Background] ECCLES JC, KOSTYUK PG, SCHMIDT RF. The effect of electric polarization of the spinal cord on central afferent fibres and on their excitatory synaptic action. J Physiol. 1962 Jun;162(1):138-50. doi: 10.1113/jphysiol.1962.sp006920. No abstract available. PMID 13889056
- [Background] Yang F, Xu Q, Cheong YK, Shechter R, Sdrulla A, He SQ, Tiwari V, Dong X, Wacnik PW, Meyer R, Raja SN, Guan Y. Comparison of intensity-dependent inhibition of spinal wide-dynamic range neurons by dorsal column and peripheral nerve stimulation in a rat model of neuropathic pain. Eur J Pain. 2014 Aug;18(7):978-88. doi: 10.1002/j.1532-2149.2013.00443.x. Epub 2014 Jan 6. PMID 24390782
- [Background] Hounsgaard J, Hultborn H, Jespersen B, Kiehn O. Bistability of alpha-motoneurones in the decerebrate cat and in the acute spinal cat after intravenous 5-hydroxytryptophan. J Physiol. 1988 Nov;405:345-67. doi: 10.1113/jphysiol.1988.sp017336. PMID 3267153
- [Background] Knikou M. Neurophysiological characterization of transpinal evoked potentials in human leg muscles. Bioelectromagnetics. 2013 Dec;34(8):630-40. doi: 10.1002/bem.21808. Epub 2013 Sep 20. PMID 24115026
- [Background] Knikou M, Dixon L, Santora D, Ibrahim MM. Transspinal constant-current long-lasting stimulation: a new method to induce cortical and corticospinal plasticity. J Neurophysiol. 2015 Sep;114(3):1486-99. doi: 10.1152/jn.00449.2015. Epub 2015 Jun 24. PMID 26108955
- [Background] Murray LM, Knikou M. Transspinal stimulation increases motoneuron output of multiple segments in human spinal cord injury. PLoS One. 2019 Mar 7;14(3):e0213696. doi: 10.1371/journal.pone.0213696. eCollection 2019. PMID 30845251
- [Background] Chen R, Tam A, Butefisch C, Corwell B, Ziemann U, Rothwell JC, Cohen LG. Intracortical inhibition and facilitation in different representations of the human motor cortex. J Neurophysiol. 1998 Dec;80(6):2870-81. doi: 10.1152/jn.1998.80.6.2870. PMID 9862891
- [Background] Devanne H, Lavoie BA, Capaday C. Input-output properties and gain changes in the human corticospinal pathway. Exp Brain Res. 1997 Apr;114(2):329-38. doi: 10.1007/pl00005641. PMID 9166922
- [Background] Bennett MR. The concept of long term potentiation of transmission at synapses. Prog Neurobiol. 2000 Feb;60(2):109-37. doi: 10.1016/s0301-0082(99)00006-4. PMID 10639051
- [Background] Sadlaoud K, Tazerart S, Brocard C, Jean-Xavier C, Portalier P, Brocard F, Vinay L, Bras H. Differential plasticity of the GABAergic and glycinergic synaptic transmission to rat lumbar motoneurons after spinal cord injury. J Neurosci. 2010 Mar 3;30(9):3358-69. doi: 10.1523/JNEUROSCI.6310-09.2010. PMID 20203195
- [Background] Ichiyama RM, Broman J, Roy RR, Zhong H, Edgerton VR, Havton LA. Locomotor training maintains normal inhibitory influence on both alpha- and gamma-motoneurons after neonatal spinal cord transection. J Neurosci. 2011 Jan 5;31(1):26-33. doi: 10.1523/JNEUROSCI.6433-09.2011. PMID 21209186
- [Background] Rossignol S, Frigon A. Recovery of locomotion after spinal cord injury: some facts and mechanisms. Annu Rev Neurosci. 2011;34:413-40. doi: 10.1146/annurev-neuro-061010-113746. PMID 21469957
- [Background] Petruska JC, Ichiyama RM, Jindrich DL, Crown ED, Tansey KE, Roy RR, Edgerton VR, Mendell LM. Changes in motoneuron properties and synaptic inputs related to step training after spinal cord transection in rats. J Neurosci. 2007 Apr 18;27(16):4460-71. doi: 10.1523/JNEUROSCI.2302-06.2007. PMID 17442831
- [Background] Ilha J, Centenaro LA, Broetto Cunha N, de Souza DF, Jaeger M, do Nascimento PS, Kolling J, Ben J, Marcuzzo S, Wyse AT, Gottfried C, Achaval M. The beneficial effects of treadmill step training on activity-dependent synaptic and cellular plasticity markers after complete spinal cord injury. Neurochem Res. 2011 Jun;36(6):1046-55. doi: 10.1007/s11064-011-0446-x. Epub 2011 Mar 22. PMID 21424738
- [Background] Ackerley SJ, Byblow WD, Barber PA, MacDonald H, McIntyre-Robinson A, Stinear CM. Primed Physical Therapy Enhances Recovery of Upper Limb Function in Chronic Stroke Patients. Neurorehabil Neural Repair. 2016 May;30(4):339-48. doi: 10.1177/1545968315595285. Epub 2015 Jul 15. PMID 26180053
- [Background] Platz T, Adler-Wiebe M, Roschka S, Lotze M. Enhancement of motor learning by focal intermittent theta burst stimulation (iTBS) of either the primary motor (M1) or somatosensory area (S1) in healthy human subjects. Restor Neurol Neurosci. 2018;36(1):117-130. doi: 10.3233/RNN-170774. PMID 29439364
- [Background] Danner SM, Hofstoetter US, Freundl B, Binder H, Mayr W, Rattay F, Minassian K. Human spinal locomotor control is based on flexibly organized burst generators. Brain. 2015 Mar;138(Pt 3):577-88. doi: 10.1093/brain/awu372. Epub 2015 Jan 12. PMID 25582580
- [Background] Ardestani MM, Henderson CE, Salehi SH, Mahtani GB, Schmit BD, Hornby TG. Kinematic and Neuromuscular Adaptations in Incomplete Spinal Cord Injury after High- versus Low-Intensity Locomotor Training. J Neurotrauma. 2019 Jun 15;36(12):2036-2044. doi: 10.1089/neu.2018.5900. Epub 2019 Feb 1. PMID 30362878
- [Background] Morrison SA, Lorenz D, Eskay CP, Forrest GF, Basso DM. Longitudinal Recovery and Reduced Costs After 120 Sessions of Locomotor Training for Motor Incomplete Spinal Cord Injury. Arch Phys Med Rehabil. 2018 Mar;99(3):555-562. doi: 10.1016/j.apmr.2017.10.003. Epub 2017 Oct 26. PMID 29107040
- [Background] Winter DA, Patla AE, Prince F, Ishac M, Gielo-Perczak K. Stiffness control of balance in quiet standing. J Neurophysiol. 1998 Sep;80(3):1211-21. doi: 10.1152/jn.1998.80.3.1211. PMID 9744933
- [Background] Sasagawa S, Ushiyama J, Masani K, Kouzaki M, Kanehisa H. Balance control under different passive contributions of the ankle extensors: quiet standing on inclined surfaces. Exp Brain Res. 2009 Jul;196(4):537-44. doi: 10.1007/s00221-009-1876-4. Epub 2009 Jun 9. PMID 19506843
- [Background] Knikou M. Function of group IB inhibition during assisted stepping in human spinal cord injury. J Clin Neurophysiol. 2012 Jun;29(3):271-7. doi: 10.1097/WNP.0b013e318257c2b7. PMID 22659724
- [Background] Desroches G, Gagnon D, Nadeau S, Popovic M. Magnitude of forward trunk flexion influences upper limb muscular efforts and dynamic postural stability requirements during sitting pivot transfers in individuals with spinal cord injury. J Electromyogr Kinesiol. 2013 Dec;23(6):1325-33. doi: 10.1016/j.jelekin.2013.09.003. Epub 2013 Sep 20. PMID 24094473
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Formento E, Minassian K, Wagner F, Mignardot JB, Le Goff-Mignardot CG, Rowald A, Bloch J, Micera S, Capogrosso M, Courtine G. Electrical spinal cord stimulation must preserve proprioception to enable locomotion in humans with spinal cord injury. Nat Neurosci. 2018 Dec;21(12):1728-1741. doi: 10.1038/s41593-018-0262-6. Epub 2018 Oct 31. PMID 30382196
- [Background] Molnar E. Long-term potentiation in cultured hippocampal neurons. Semin Cell Dev Biol. 2011 Jul;22(5):506-13. doi: 10.1016/j.semcdb.2011.07.017. Epub 2011 Jul 22. PMID 21807105
- [Background] Kobayashi M, Pascual-Leone A. Transcranial magnetic stimulation in neurology. Lancet Neurol. 2003 Mar;2(3):145-56. doi: 10.1016/s1474-4422(03)00321-1. PMID 12849236
- [Background] Dixon L, Ibrahim MM, Santora D, Knikou M. Paired associative transspinal and transcortical stimulation produces plasticity in human cortical and spinal neuronal circuits. J Neurophysiol. 2016 Aug 1;116(2):904-16. doi: 10.1152/jn.00259.2016. Epub 2016 Jun 8. PMID 27281748
- [Background] Hanna-Boutros B, Sangari S, Giboin LS, El Mendili MM, Lackmy-Vallee A, Marchand-Pauvert V, Knikou M. Corticospinal and reciprocal inhibition actions on human soleus motoneuron activity during standing and walking. Physiol Rep. 2015 Feb 25;3(2):e12276. doi: 10.14814/phy2.12276. PMID 25825912
- [Background] Hannah R, Cavanagh SE, Tremblay S, Simeoni S, Rothwell JC. Selective Suppression of Local Interneuron Circuits in Human Motor Cortex Contributes to Movement Preparation. J Neurosci. 2018 Jan 31;38(5):1264-1276. doi: 10.1523/JNEUROSCI.2869-17.2017. Epub 2017 Dec 20. PMID 29263237
- [Background] Alexeeva N, Broton JG, Calancie B. Latency of changes in spinal motoneuron excitability evoked by transcranial magnetic brain stimulation in spinal cord injured individuals. Electroencephalogr Clin Neurophysiol. 1998 Aug;109(4):297-303. doi: 10.1016/s0924-980x(98)00021-6. PMID 9751291
- [Background] Geertsen SS, Zuur AT, Nielsen JB. Voluntary activation of ankle muscles is accompanied by subcortical facilitation of their antagonists. J Physiol. 2010 Jul 1;588(Pt 13):2391-402. doi: 10.1113/jphysiol.2010.190678. Epub 2010 May 10. PMID 20457734
- [Background] Dobkin B, Apple D, Barbeau H, Basso M, Behrman A, Deforge D, Ditunno J, Dudley G, Elashoff R, Fugate L, Harkema S, Saulino M, Scott M; Spinal Cord Injury Locomotor Trial Group. Weight-supported treadmill vs over-ground training for walking after acute incomplete SCI. Neurology. 2006 Feb 28;66(4):484-93. doi: 10.1212/01.wnl.0000202600.72018.39. PMID 16505299
- [Background] Roby-Brami A, Bussel B. Long-latency spinal reflex in man after flexor reflex afferent stimulation. Brain. 1987 Jun;110 ( Pt 3):707-25. doi: 10.1093/brain/110.3.707. PMID 3107749
- [Background] Grey MJ, Klinge K, Crone C, Lorentzen J, Biering-Sorensen F, Ravnborg M, Nielsen JB. Post-activation depression of soleus stretch reflexes in healthy and spastic humans. Exp Brain Res. 2008 Feb;185(2):189-97. doi: 10.1007/s00221-007-1142-6. Epub 2007 Oct 12. PMID 17932663
- [Background] Schindler-Ivens S, Shields RK. Low frequency depression of H-reflexes in humans with acute and chronic spinal-cord injury. Exp Brain Res. 2000 Jul;133(2):233-41. doi: 10.1007/s002210000377. PMID 10968224
- [Background] Thompson AK, Wolpaw JR. Operant conditioning of spinal reflexes: from basic science to clinical therapy. Front Integr Neurosci. 2014 Mar 18;8:25. doi: 10.3389/fnint.2014.00025. eCollection 2014. PMID 24672441
- [Background] Thompson AK, Wolpaw JR. Restoring walking after spinal cord injury: operant conditioning of spinal reflexes can help. Neuroscientist. 2015 Apr;21(2):203-15. doi: 10.1177/1073858414527541. Epub 2014 Mar 17. PMID 24636954
- [Background] Thompson AK, Pomerantz FR, Wolpaw JR. Operant conditioning of a spinal reflex can improve locomotion after spinal cord injury in humans. J Neurosci. 2013 Feb 6;33(6):2365-75. doi: 10.1523/JNEUROSCI.3968-12.2013. PMID 23392666
- [Background] Crone C, Nielsen J. Methodological implications of the post activation depression of the soleus H-reflex in man. Exp Brain Res. 1989;78(1):28-32. doi: 10.1007/BF00230683. PMID 2591515
- [Background] Aymard C, Katz R, Lafitte C, Lo E, Penicaud A, Pradat-Diehl P, Raoul S. Presynaptic inhibition and homosynaptic depression: a comparison between lower and upper limbs in normal human subjects and patients with hemiplegia. Brain. 2000 Aug;123 ( Pt 8):1688-702. doi: 10.1093/brain/123.8.1688. PMID 10908198
- [Background] Crone C, Hultborn H, Jespersen B, Nielsen J. Reciprocal Ia inhibition between ankle flexors and extensors in man. J Physiol. 1987 Aug;389:163-85. doi: 10.1113/jphysiol.1987.sp016652. PMID 3681725
- [Background] Mummidisetty CK, Smith AC, Knikou M. Modulation of reciprocal and presynaptic inhibition during robotic-assisted stepping in humans. Clin Neurophysiol. 2013 Mar;124(3):557-64. doi: 10.1016/j.clinph.2012.09.007. Epub 2012 Oct 6. PMID 23046639
- [Background] Simonsen EB, Dyhre-Poulsen P. Amplitude of the human soleus H reflex during walking and running. J Physiol. 1999 Mar 15;515 ( Pt 3)(Pt 3):929-39. doi: 10.1111/j.1469-7793.1999.929ab.x. PMID 10066917
- [Background] Smith AC, Knikou M. A Review on Locomotor Training after Spinal Cord Injury: Reorganization of Spinal Neuronal Circuits and Recovery of Motor Function. Neural Plast. 2016;2016:1216258. doi: 10.1155/2016/1216258. Epub 2016 May 11. PMID 27293901
- [Background] Knikou M. The H-reflex as a probe: pathways and pitfalls. J Neurosci Methods. 2008 Jun 15;171(1):1-12. doi: 10.1016/j.jneumeth.2008.02.012. Epub 2008 Mar 4. PMID 18394711
- [Background] Bethoux F, Bennett S. Evaluating walking in patients with multiple sclerosis: which assessment tools are useful in clinical practice? Int J MS Care. 2011 Spring;13(1):4-14. doi: 10.7224/1537-2073-13.1.4. PMID 24453700
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Learmonth YC, Paul L, McFadyen AK, Mattison P, Miller L. Reliability and clinical significance of mobility and balance assessments in multiple sclerosis. Int J Rehabil Res. 2012 Mar;35(1):69-74. doi: 10.1097/MRR.0b013e328350b65f. PMID 22315143
- [Background] Behrman AL, Ardolino EM, Harkema SJ. Activity-Based Therapy: From Basic Science to Clinical Application for Recovery After Spinal Cord Injury. J Neurol Phys Ther. 2017 Jul;41 Suppl 3(Suppl 3 IV STEP Spec Iss):S39-S45. doi: 10.1097/NPT.0000000000000184. PMID 28628595
- [Background] Kirshblum SC, Burns SP, Biering-Sorensen F, Donovan W, Graves DE, Jha A, Johansen M, Jones L, Krassioukov A, Mulcahey MJ, Schmidt-Read M, Waring W. International standards for neurological classification of spinal cord injury (revised 2011). J Spinal Cord Med. 2011 Nov;34(6):535-46. doi: 10.1179/204577211X13207446293695. No abstract available. PMID 22330108
- [Background] Zorner B, Blanckenhorn WU, Dietz V; EM-SCI Study Group; Curt A. Clinical algorithm for improved prediction of ambulation and patient stratification after incomplete spinal cord injury. J Neurotrauma. 2010 Jan;27(1):241-52. doi: 10.1089/neu.2009.0901. PMID 19645527
- [Background] Kraemer HC. A Source of False Findings in Published Research Studies: Adjusting for Covariates. JAMA Psychiatry. 2015 Oct;72(10):961-2. doi: 10.1001/jamapsychiatry.2015.1178. No abstract available. PMID 26244634
- [Background] van Middendorp JJ, Hosman AJ, Pouw MH; EM-SCI Study Group; Van de Meent H. ASIA impairment scale conversion in traumatic SCI: is it related with the ability to walk? A descriptive comparison with functional ambulation outcome measures in 273 patients. Spinal Cord. 2009 Jul;47(7):555-60. doi: 10.1038/sc.2008.162. Epub 2008 Dec 23. PMID 19104512
- [Background] van Middendorp JJ, Hosman AJ, Donders AR, Pouw MH, Ditunno JF Jr, Curt A, Geurts AC, Van de Meent H; EM-SCI Study Group. A clinical prediction rule for ambulation outcomes after traumatic spinal cord injury: a longitudinal cohort study. Lancet. 2011 Mar 19;377(9770):1004-10. doi: 10.1016/S0140-6736(10)62276-3. Epub 2011 Mar 4. PMID 21377202
- [Background] Dong Y, Peng CY. Principled missing data methods for researchers. Springerplus. 2013 May 14;2(1):222. doi: 10.1186/2193-1801-2-222. Print 2013 Dec. PMID 23853744
- [Derived] Skiadopoulos A, Famodimu GO, Solomon SK, Agarwal P, Harel NY, Knikou M. Priming locomotor training with transspinal stimulation in people with spinal cord injury: study protocol of a randomized clinical trial. Trials. 2023 Feb 25;24(1):145. doi: 10.1186/s13063-023-07193-4. PMID 36841773
- [Derived] Skiadopoulos A, Famodimu GO, Solomon SK, Agrawal P, Harel NY, Knikou M. Priming locomotor training with transspinal stimulation in people with spinal cord injury: study protocol of a randomized clinical trial. Res Sq [Preprint]. 2023 Feb 16:rs.3.rs-2527617. doi: 10.21203/rs.3.rs-2527617/v1. PMID 36824823